CLINICAL TRIAL: NCT05729542
Title: Randomized Controlled Trial Comparing Clinical Outcomes of Patients Treated Surgically With Suture Button Versus Fibulink Fixation for Acute Ankle Syndesmosis Injuries
Brief Title: Comparing Clinical Outcomes of Suture Button Versus Fibulink Fixation for Acute Ankle Syndesmosis Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, William Kent, Assistant Professor of Orthopaedic Surgery, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 800669
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ankle Injuries; Syndesmotic Injuries; Ankle Fractures
MeSH Terms: conditions — Ankle Injuries; Ankle Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arthrex Tightrope (Active Comparator): Syndesmosis fixation performed with ARthrex Tightrope device. This is a high-tension suture fixation with a button based anchor system.
  Interventions: Device: Arthrex Tightrope
- Synthes Fibulink (Experimental): Syndesmosis fixation perforemd with Synthes Fibulink device. This is a high-tension fixation with a screw based anchor system.
  Interventions: Device: Synthes Fibulink

INTERVENTIONS:
Device: Arthrex Tightrope — High-tensile strength suture syndesmosis repair
  Arms: Arthrex Tightrope
Device: Synthes Fibulink — High-tensile strength suture syndesmosis repair
  Arms: Synthes Fibulink

SUMMARY:
This project consists of a randomized controlled study design. Study candidates will include all patients 18 years or older, who were evaluated at UCSD and found to have an acute ankle syndesmosis injury requiring surgery. Patients who consent to study participation will be randomized to receive one of two standard of care procedures - either a suture button or Fibulink implant. Outcome measures, including the Olerud-Molander and American Orthopaedic Foot and Ankle Society scores, pain, range of motion, time to return to work, and radiographic evaluation will be collected for each participant. Given the potential degenerative changes and poor radiographic and clinical outcomes with inadequate repair of the syndesmosis, it is imperative to evaluate existing and emerging methods of fixation for patients with acute ankle fractures with syndesmosis injuries.

ELIGIBILITY:
Inclusion Criteria:

* Ankle fracture with associated syndesmotic injury requiring surgery
* Age 18 years or older
* Ability to understand the content of the patient information/informed consent form

Exclusion Criteria:

* Any not medically managed severe systemic disease
* Patient preference for specific implant
* Refusal of randomization
* Pregnant patients
* Prisoners
* Participation in any other pharmacologic or medicinal product study within the previous month that could influence the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Pain score | 1 year
  VAS Pain score is rated from 0-10, 0=no pain and 10=most severe pain
Foot and Ankle Disability Index | 1 year
  Functional score with a 0-104 with higher scores indicating better function
Olerud-Molander Ankle Score | 1 year
  Functional Score with a score of 0-100 with higher scores indicating better function

SECONDARY OUTCOMES:
Number of participants with medical or surgical complications | 1 year
  Medical and surgical complications to include: surgical site infection, re-operation, device failure, loss of motion

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No